CLINICAL TRIAL: NCT03529461
Title: Use of Non-Invasive Positive Pressure Ventilation in Patients With Severe Obesity Undergoing Upper Endoscopy Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol Hospital (Other)
Responsible Party: Principal Investigator, Makram Gedeon, MD, Medical director of bariatric surgery program, principal investigator, Bristol Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20170730
Record Dates: First submitted 2018-05-03; First posted 2018-05-18 (Actual); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Severe Obesity; Hypoxia
Keywords: severe obesity; non-invasive positive pressure ventilation; endoscopy; hypoxia; bariatric surgery; sedation; adverse events; BMI; anesthesia; complications
MeSH Terms: conditions — Obesity, Morbid; Hypoxia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Other): Intervention: nasal cannula (6L O2) + non invasive positive pressure nasal mask (not connected to machine)
  Interventions: Device: Rescue non-invasive positive pressure ventilation through nasal mask; Other: Secondary rescue maneuvers
- Experimental (Experimental): Intervention: Non invasive positive pressure nasal mask (connect to machine once patient is sedated)
  Interventions: Device: Non-invasive positive pressure ventilation through nasal mask; Other: Secondary rescue maneuvers

INTERVENTIONS:
Device: Non-invasive positive pressure ventilation through nasal mask — Inspiratory pressure 12 cm H2O/Expiratory pressure 6 cm H2O which can be increased to meet a tidal volume (TV) of 300-800 mL (target is 450-500), with maximum Inspiratory pressure 18 cm H2O /Expiratory pressure 8 cm H2O on 100% FiO2.If TVs are more or less than 300 to 800 mL range, the pressure will be adjusted by 1-2 cm H2O) accordingly
  Arms: Experimental
Device: Rescue non-invasive positive pressure ventilation through nasal mask — If desaturation below 90 %, nasal cannula removed and non invasive positive pressure nasal mask connected to machine: Inspiratory pressure 12 cm H2O/Expiratory pressure 6 cm H2O which can be increased to meet a tidal volume (TV) of 300-800 mL (target is 450-500), with maximum Inspiratory pressure 18 cm H2O /Expiratory pressure 8 cm H2O on 100% FiO2.If TVs are more or less than 300 to 800 mL range, the pressure will be adjusted by 1-2 cm H2O) accordingly
  Arms: Control
Other: Secondary rescue maneuvers — If rescue non invasive positive pressure maneuver attempted (including adjustments in pressure) and O2 sat is not above 90 % within 3 min of starting non invasive positive pressure, scope removed and secondary rescue maneuver started. Secondary rescue maneuvers performed at the discretion of the anesthesiologist (chin lift, oral airway, bag mask, nasal trumpet, LMA, intubation). If sat > 90 % with secondary rescue maneuvers, resumption of scope exam to the discretion of anesthesia. If sat does not increase > 90 % with secondary rescue maneuvers, scope exam to be cancelled and patient care per anesthesiologist

SUMMARY:
The study evaluated the effect of non-invasive positive pressure ventilation (NIPPV) to decrease the incidence of desaturation events in patients with severe obesity undergoing upper endoscopy.

DETAILED DESCRIPTION:
Patients being evaluated for bariatric surgery often undergo preoperative upper endoscopy. Patients with obesity are at increased risk for sedation related adverse events during endoscopy. The study evaluated the effect of non-invasive positive pressure ventilation (NIPPV) to decrease the incidence of desaturation in patients with severe obesity undergoing upper endoscopy. The study was a randomized controlled trial that assessed the effectiveness of NIPPV in patients undergoing upper endoscopy. Patients were randomized into experimental group NIPPV or control group. Primary endpoints were desaturation events (SpO2 <=94%) and desaturation events requiring intervention (SpO2<=90%). A secondary endpoint was the use of NIPPV to rescue patients who developed a clinically significant desaturation event.

ELIGIBILITY:
Inclusion Criteria:

* Weight loss surgery patients undergoing preoperative upper endoscopy
* BMI 40-60

Exclusion Criteria:

* Pregnant patients
* Previous weight loss surgery or stomach surgery
* BMI > 60 and BMI < 40
* Active smokers
* Patients with a history of recent URTI (Upper Respiratory Tract Infection) within the preceding 2 weeks
* Lung disease, COPD asthma, cystic fibrosis, sarcoidosis
* Baseline O2 saturation less than or equal to 94%
* Exclude substance abusers (active alcohol abuse, benzodiazepine abuse, and active illicit drug use)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Makram M Gedeon, MD, Principal Investigator — Bristol Hospital
Locations (1):
- Bristol Hospital, Bristol, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross JB, Bachenberg KL, Benumof JL, Caplan RA, Connis RT, Cote CJ, Nickinovich DG, Prachand V, Ward DS, Weaver EM, Ydens L, Yu S; American Society of Anesthesiologists Task Force on Perioperative Management. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: a report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2006 May;104(5):1081-93; quiz 1117-8. doi: 10.1097/00000542-200605000-00026. No abstract available. PMID 16645462
- [Background] Arakawa H, Kaise M, Sumiyama K, Saito S, Suzuki T, Tajiri H. Does pulse oximetry accurately monitor a patient's ventilation during sedated endoscopy under oxygen supplementation? Singapore Med J. 2013 Apr;54(4):212-5. doi: 10.11622/smedj.2013075. PMID 23624448
- [Background] De Palma GD, Forestieri P. Role of endoscopy in the bariatric surgery of patients. World J Gastroenterol. 2014 Jun 28;20(24):7777-84. doi: 10.3748/wjg.v20.i24.7777. PMID 24976715
- [Background] Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91. doi: 10.1001/jama.2016.6458. PMID 27272580
- [Background] Fouladpour N, Jesudoss R, Bolden N, Shaman Z, Auckley D. Perioperative Complications in Obstructive Sleep Apnea Patients Undergoing Surgery: A Review of the Legal Literature. Anesth Analg. 2016 Jan;122(1):145-51. doi: 10.1213/ANE.0000000000000841. PMID 26111263
- [Background] Gay PC. Complications of noninvasive ventilation in acute care. Respir Care. 2009 Feb;54(2):246-57; discussion 257-8. PMID 19173756
- [Background] Gomez V, Bhalla R, Heckman MG, Florit PT, Diehl NN, Rawal B, Lynch SA, Loeb DS. Routine Screening Endoscopy before Bariatric Surgery: Is It Necessary? Bariatr Surg Pract Patient Care. 2014 Dec 1;9(4):143-149. doi: 10.1089/bari.2014.0024. PMID 25516819
- [Background] Goudra BG, Singh PM, Penugonda LC, Speck RM, Sinha AC. Significantly reduced hypoxemic events in morbidly obese patients undergoing gastrointestinal endoscopy: Predictors and practice effect. J Anaesthesiol Clin Pharmacol. 2014 Jan;30(1):71-7. doi: 10.4103/0970-9185.125707. PMID 24574597
- [Background] McVay T, Fang JC, Taylor L, Au A, Williams W, Presson AP, Al-Dulaimi R, Volckmann E, Ibele A. Safety Analysis of Bariatric Patients Undergoing Outpatient Upper Endoscopy with Non-Anesthesia Administered Propofol Sedation. Obes Surg. 2017 Jun;27(6):1501-1507. doi: 10.1007/s11695-016-2478-4. PMID 27885537
- [Background] Opperer M, Cozowicz C, Bugada D, Mokhlesi B, Kaw R, Auckley D, Chung F, Memtsoudis SG. Does Obstructive Sleep Apnea Influence Perioperative Outcome? A Qualitative Systematic Review for the Society of Anesthesia and Sleep Medicine Task Force on Preoperative Preparation of Patients with Sleep-Disordered Breathing. Anesth Analg. 2016 May;122(5):1321-34. doi: 10.1213/ANE.0000000000001178. PMID 27101493
- [Background] Saunders R, Erslon M, Vargo J. Modeling the costs and benefits of capnography monitoring during procedural sedation for gastrointestinal endoscopy. Endosc Int Open. 2016 Mar;4(3):E340-51. doi: 10.1055/s-0042-100719. PMID 27004254
- [Background] Slagelse C, Vilmann P, Hornslet P, Jorgensen HL, Horsted TI. The role of capnography in endoscopy patients undergoing nurse-administered propofol sedation: a randomized study. Scand J Gastroenterol. 2013 Oct;48(10):1222-30. doi: 10.3109/00365521.2013.830327. Epub 2013 Sep 2. PMID 23992025
- [Background] Soto RG, Davis M, Faulkner MJ. A comparison of the incidence of hypercapnea in non-obese and morbidly obese peri-operative patients using the SenTec transcutaneous pCO(2) monitor. J Clin Monit Comput. 2014 Jun;28(3):293-8. doi: 10.1007/s10877-013-9534-6. Epub 2013 Nov 29. PMID 24292821
- [Background] Wani S, Azar R, Hovis CE, Hovis RM, Cote GA, Hall M, Waldbaum L, Kushnir V, Early D, Mullady DK, Murad F, Edmundowicz SA, Jonnalagadda SS. Obesity as a risk factor for sedation-related complications during propofol-mediated sedation for advanced endoscopic procedures. Gastrointest Endosc. 2011 Dec;74(6):1238-47. doi: 10.1016/j.gie.2011.09.006. PMID 22136773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 4/25/2017 and ended on 4/2/2018.
Pre-assignment Details: 208 patients assessed for eligibility:
  * 56 patients enrolled
  * 152 patients excluded (reasons: 127 not meeting inclusion criteria or no show for procedure, 6 patients declined to participate, 19 patients excluded because of early trial closure)
Groups:
- Control: Intervention: nasal cannula 6L O2 + non invasive positive pressure (NIPPV) nasal mask not connected to machine
  Rescue NIPPV via nasal mask: If oxygen desaturation below 90 %. IPAP 12 cm H2O/EPAP 6 cm H2O titrated to meet a tidal volume of 300-800mL target is 450-500, with maximum IPAP 18cm H2O /EPAP 8 cm H2O on 100% FiO2.If TVs are more or less than 300 to 800 mL range the pressure will be adjusted by 1-2 cm H2O.
  Secondary rescue maneuvers: If rescue non invasive positive pressure maneuver attempted and O2 saturation is not above 90 % within 3 min of starting non invasive positive pressure, scope removed and secondary rescue maneuver started. Secondary rescue maneuvers performed at the discretion of the anesthesiologist. If oxygen saturation > 94 % with secondary rescue maneuvers, resumption of scope exam to the discretion of anesthesia. If saturation does not increase > 94 % with secondary rescue maneuvers, scope exam cancelled and patient care per anesthesiologist
- Experimental: Intervention: NIPP placed on patient. Positive pressure applied once patient is sedated
  NIPPV through nasal mask: IPAP 12cm H2O/EPAP 6cm H2O titrated to tidal volume of 300-800 mL (target 450-500), maximum IPAP 18 cm H2O /EPAP 8 cm H2O on 100% FiO2.If TVs are more or less than 300 to 800 mL range, pressure will be adjusted by 1-2 cm H2O.
  Secondary rescue maneuvers: If rescue NIPPV maneuver attempted (including adjustments in pressure) and O2 saturation is not above 90 % within 3 min of starting NIPPV, endoscope removed and secondary rescue maneuver started. Secondary rescue maneuvers performed at the discretion of the anesthesiologist (chin lift, oral airway, bag mask, nasal trumpet, LMA, intubation). If saturation > 94 % with secondary rescue maneuvers, resumption of scope exam to the discretion of anesthesia. If saturation does not increase > 94 % with secondary rescue maneuvers, scope exam to be cancelled and patient care per anesthesiologist
Period: Overall Study
Arm/Group | Control | Experimental
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Intervention: nasal cannula 6L O2 + non invasive positive pressure nasal mask not connected to machine
  Rescue NIPPV via nasal mask: If desaturation below 90 %. IPAP 12 cm H2O/EPAP 6 cm H2O titrated to meet a tidal volume of 300-800mL target is 450-500, with maximum IPAP 18cm H2O /EPAP 8 cm H2O on 100% FiO2.If TVs are more or less than 300 to 800 mL range the pressure will be adjusted by 1-2 cm H2O.
  Secondary rescue maneuvers: If rescue non invasive positive pressure maneuver attempted and O2 sat is not above 90 % within 3 min of starting non invasive positive pressure, scope removed and secondary rescue maneuver started. Secondary rescue maneuvers performed at the discretion of the anesthesiologist. If sat > 94 % with secondary rescue maneuvers, resumption of scope exam to the discretion of anesthesia. If sat does not increase > 94 % with secondary rescue maneuvers, scope exam cancelled and patient care per anesthesiologist
- Experimental: Intervention: Non invasive positive pressure nasal mask connected once patient is sedated
  NIPPV through nasal mask: IPAP 12cm H2O/EPAP 6cm H2O titrated to tidal volume of 300-800 mL (target 450-500), maximum IPAP 18 cm H2O /EPAP 8 cm H2O on 100% FiO2.If TVs are more or less than 300 to 800 mL range, pressure will be adjusted by 1-2 cm H2O.
  Secondary rescue maneuvers: If rescue non invasive positive pressure maneuver attempted (including adjustments in pressure) and O2 sat is not above 90 % within 3 min of starting non invasive positive pressure, scope removed and secondary rescue maneuver started. Secondary rescue maneuvers performed at the discretion of the anesthesiologist (chin lift, oral airway, bag mask, nasal trumpet, LMA, intubation). If sat > 94 % with secondary rescue maneuvers, resumption of scope exam to the discretion of anesthesia. If sat does not increase > 94 % with secondary rescue maneuvers, scope exam to be cancelled and patient care per anesthesiologist
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (11.6) | 36.5 (11.8) | 37.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Oxygen Desaturation Event ≤ 94%
Description: Percentage of participants who develop a peripheral oxygen saturation measured by pulse oximetry ≤ 94%
Time Frame: Time in seconds beginning with the start of procedure (anesthesia induction) ending with procedure completion (eyes open to verbal stimuli).
Measure: Number; unit: percentage of participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 28 | 28
percentage of participants | 57.1 | 14.3

2. Primary Outcome: Percentage of Participants With an Oxygen Desaturation Event < 90%
Description: Percentage of participants who develop a peripheral oxygen saturation event < 90%.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 28 | 28
percentage of participants | 28.6 | 3.5

3. Secondary Outcome: Percentage of Participants in the Control Group With an Oxygen Saturation Less Than 90 % Who Responded to Rescue NIPPV
Description: We used non-invasive positive pressure ventilation (NIPPV) as a first rescue maneuver in control patients who developed an oxygen desaturation less than 90 % and reported on the percentage of participants who responded. The rescue was considered successful with recovery of oxygen saturation more than 90 % within 3 minutes.
Time Frame: 3 minutes following a desaturation event < 90 %
Population: We report on the response of 8 participants in the control group who had an oxygen desaturation event less than 90 %
Measure: Count of Participants; unit: Participants
Groups:
- Control Participants With Oxygen Desaturation < 90%: Rescue NIPPV: If desaturation below 90 %. IPAP 12 cm H2O/EPAP 6 cm H2O titrated to meet a tidal volume of 300-800mL target is 450-500, with maximum IPAP 18cm H2O /EPAP 8 cm H2O on 100% FiO2.If TVs are more or less than 300 to 800 mL range the pressure will be adjusted by 1-2 cm H2O. If rescue non invasive positive pressure maneuver attempted and O2 sat is not above 90 % within 3 min of starting non invasive positive pressure, scope removed and secondary rescue maneuver started. Secondary rescue maneuvers performed at the discretion of the anesthesiologist. If sat > 94 % with secondary rescue maneuvers, resumption of scope exam to the discretion of anesthesia. If sat does not increase > 94 % with secondary rescue maneuvers, scope exam cancelled and patient care per anesthesiologist
Arm/Group | Control Participants With Oxygen Desaturation < 90%
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 1800 seconds (30 minutes)
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT03529461/Prot_SAP_ICF_001.pdf